CLINICAL TRIAL: NCT02071849
Title: HAART 200 Aortic Valve Annuloplasty During Bicuspid Aortic Valve Reconstruction Trial
Brief Title: HAART 200 Aortic Valve Annuloplasty Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biostable Science & Engineering (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-01-025
Record Dates: First submitted 2014-02-17; First posted 2014-02-26 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Aortic Insufficiency
Keywords: Aortic Insufficiency; Aortic Regurgitation
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aortic Valve Repair (Experimental): Implantation of HAART 200 Aortic Valve Annuloplasty Device for bicuspid aortic valve reconstruction
  Interventions: Device: HAART 200 Aortic Valve Annuloplasty Device

INTERVENTIONS:
Device: HAART 200 Aortic Valve Annuloplasty Device — Surgical repair of bicuspid aortic valve using the HAART 200 Aortic Valve Annuloplasty Device .

SUMMARY:
The HAART 200 "Aortic Annuloplasty during Bicuspid Aortic Valve Reconstruction" Trial is a prospective, non-randomized, multi-center trial to evaluate the safety and effectiveness of the HAART 200 bicuspid annuloplasty ring when used to surgically stabilize the aortic valve annulus in patients undergoing repair of bicuspid aortic valves (BAV) for predominant aortic insufficiency (AI).

DETAILED DESCRIPTION:
Aortic valve disease is the most common valvular heart disease with approximately 200,000 patients per year undergoing conventional aortic valve replacement in North America and Europe. Around 60% of valves have Aortic Stenosis (AS) and 40% of have Aortic Insufficiency, which is the failure of the aortic valve to close completely during diastole, causing blood to flow from the aorta back into the left ventricle. Bicuspid valve morphology is present in a fourth to a third of patients coming to surgical intervention, and constitutes a very important subset. Several conditions are associated with bicuspid disease, including ascending aortic or root aneurysms in up to a third.

Traditional management of aortic valve and root disease has been with aortic valve replacement, with or without root replacement (Bentall Procedure). However, as has been observed in patients with mitral valve repair, the option of maintaining one's reconstructed native valve versus a replacement, either bioprosthetic or mechanical, can have multiple benefits. The advantages of repair include: the avoidance of prosthetic valve related complications and structural degeneration with bioprosthetic valves over 10-15 years and elimination of the need for anticoagulation and related problems with mechanical valves in younger patients. The significantly lower rate of endocarditis after repair is a major impetus to increasing performance of BAV reconstruction. Thus, aortic valve repair currently is established as an excellent option for patients with BAV. However, with connective tissue disorders being an inherent feature of BAV, outcomes have been less stable long-term than for trileaflet repair, primarily because of late annular redilatation in BAV disease.

Therefore, this study is designed to evaluate the safety and effectiveness of annular stabilization with a bicuspid annuloplasty ring in patients undergoing repair of a bicuspid aortic valve for predominant aortic insufficiency.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 18 years of age or older
2. The subject has bi-leaflet aortic valve morphology
3. The subject has documented aortic valve disease which may or may not include:

   * Aortic valve insufficiency
   * Ascending aortic or aortic root pathology
   * Other pathology of the ascending aorta that requires elective aortic replacement
   * Associated stable one or two vessel coronary disease requiring concomitant coronary bypass
   * Patients with recurrent severe AI (Grade 3 or 4) after prior bicuspid repair who are undergoing re-repair because of annular re-dilatation
   * All bicuspid annular and leaflet configurations will be included
4. The subject needs:

   * correction of BAV annular dilatation in patients with chronic AI and dilated annulus
   * restoration of a circular annular shape in patients with bicuspid valve and expansion of sinus to sinus dimensions
   * stabilization of annular geometry long-term in rare bicuspid valve patients with severe AI and minimal annular dilatation
5. The is willing to comply with specified follow-up evaluations, including transesophageal echocardiography (TEE) if there are inadequate images by transthoracic echocardiography (TTE) to assess the aortic valve
6. The subject has reviewed and signed the written informed consent form
7. The subject agrees to return for all follow-up evaluations for the duration of the study (i.e. geographically stable)

Exclusion Criteria:

1. All patients will be excluded who require emergency surgery for any reason.
2. All the patients who have had a prior heart valve replacement
3. The subject's aortic valve morphology is not bicuspid.
4. The subject has active endocarditis
5. The subject has mixed stenosis and regurgitation of the aortic valve with predominant stenosis
6. Heavily calcified BAV valves, calcified aortic roots, or "porcelain aortas"
7. Leukopenia with a White Blood Cell (WBC) of less than 3000
8. Acute anemia with a Hgb less than 9mg%
9. Platelet count less than 100,000 cells/mm3
10. History of a defined bleeding diathesis or coagulopathy or the subject refuses blood transfusions
11. Active infection requiring antibiotic therapy (if temporary illness, subjects may enroll 2-4 weeks after discontinuation of antibiotics)
12. Subjects in whom transesophageal echocardiography (TEE) is contraindicated
13. Low Ejection Fraction (EF) < 35%
14. Life expectancy < 1 year, or severe comorbidities, such as dialysis or severe Chronic Obstructive Pulmonary Disease (COPD)
15. The subject is or will be participating in a concomitant research study of an investigational product or has participated in such a study within the 30 days prior to screening
16. The subject is a minor, an illicit drug user, alcohol abuser, prisoner, institutionalized, or is unable to give informed consent
17. The subject is pregnant or lactating
18. Recent (within 6 months) cerebrovascular accident (CVA) or a transient ischemic attack (TIA)
19. Myocardial Infarction (MI) within one month of trial inclusion
20. The subject has a known intolerance to titanium or polyester
21. The subject has documented unstable or > 2 vessel coronary disease
22. The subject requires additional valve replacement or valve repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominico Mazzitelli, MD, Principal Investigator — München Heart Center
Locations (4):
- Germany (4):
  - München Heart Center, München, Bavaria
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - Klinik und Poliklinik für Herz- und Gefäßchirurgie, Hamburg
  - Klinikum Nürnberg Süd, Nuremberg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mazzitelli D, Pfeiffer S, Rankin JS, Fischlein T, Choi YH, Wahlers T, Nobauer C, Schreiber C, Lange R. A Regulated Trial of Bicuspid Aortic Valve Repair Supported by Geometric Ring Annuloplasty. Ann Thorac Surg. 2015 Jun;99(6):2010-6. doi: 10.1016/j.athoracsur.2015.01.050. Epub 2015 Apr 10. PMID 25865762

RESULTS

PARTICIPANT FLOW:
Period: 6-month Primary Endpoint
Arm/Group | Aortic Valve Repair
Started | 20
Completed | 15
Not Completed | 5
Not completed — Did not receive device | 4
Not completed — Adverse Event | 1
Period: 2-year Extended Follow-up
Arm/Group | Aortic Valve Repair
Started | 15
Completed | 14
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: 16 of 20 consented participants received the device
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (11.3)
Age, Customized [Count of Participants; unit: Participants]
  18-29 | 3
  30-39 | 2
  40-49 | 6
  50-59 | 4
  60-69 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Region of Enrollment [Number; unit: participants]
  Germany | 16
Aortic Insufficiency [Count of Participants; unit: Participants] — Grade assigned to degree of aortic regurgitation determined by core laboratory analysis of echocardiogram:
  0=None/trace,1+=Mild, 2+=Moderate, 3+=Moderately Severe, 4+=Severe
  Participants
    0 | 1
    1+ | 3
    2+ | 2
    3+ | 5
    4+ | 3
    Grade not available | 2
New York Heart Association (NYHA) Functional Capacity [Count of Participants; unit: Participants] — Four classes describing the effect of cardiac disease on physical activity: Class I - disease does not limit activity; Class II - slight limitation; Class III - marked limitation; Class IV - inability to carry out any physical activity without discomfort
  Participants
    I | 3
    II | 13
    III | 0
    IV | 0
Peak gradient [Mean (Standard Deviation); unit: mm Hg] — Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  mm Hg
    number analyzed (Participants) | 13
    (all) | 25.5 (22.3)
Mean gradient [Mean (Standard Deviation); unit: mm Hg] — Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  mm Hg
    number analyzed (Participants) | 13
    (all) | 13.4 (12.9)
Left ventricular (LV) mass [Mean (Standard Deviation); unit: g] — Left ventricular mass. Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  g
    number analyzed (Participants) | 13
    (all) | 288.62 (90.23)
Left ventricular internal dimension (LVID) diastole [Mean (Standard Deviation); unit: cm] — Left ventricular internal dimension. Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  cm
    number analyzed (Participants) | 13
    (all) | 5.408 (0.952)
LVID systole [Mean (Standard Deviation); unit: cm] — Left ventricular internal dimension. Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  cm
    number analyzed (Participants) | 11
    (all) | 3.527 (0.793)
LV diastolic volume [Mean (Standard Deviation); unit: ml] — Left ventricular diastolic volume. Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  ml
    number analyzed (Participants) | 11
    (all) | 144.5 (57.6)
LV systolic volume [Mean (Standard Deviation); unit: ml] — Left ventricular systolic volume. Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  ml
    number analyzed (Participants) | 11
    (all) | 69.1 (36.6)
Left ventricular ejection fraction (LVEF) [Mean (Standard Deviation); unit: percentage of blood volume] — Left ventricular ejection fraction. Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  percentage of blood volume
    number analyzed (Participants) | 11
    (all) | 53.86 (8.76)
Cardiac output [Mean (Standard Deviation); unit: l/min] — Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  l/min
    number analyzed (Participants) | 12
    (all) | 7.926 (2.365)
Cardiac index [Mean (Standard Deviation); unit: l/min/m^2] — Cardiac index is the cardiac output divided by body surface area. Population: Participants with an echocardiogram evaluable for this measure.
  l/min/m^2
    number analyzed (Participants) | 12
    (all) | 3.88 (1.16)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Outcome Measure: Survival Defined as Survival Free From All Cause Death at 6 Months Postprocedure.
Time Frame: 6 months postprocedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 16
percentage of participants | 100 [79.4 to 100]

2. Primary Outcome: Primary Efficacy Outcome Measure: Aortic Insufficiency (AI) at 6 Months
Description: Aortic insufficiency assessed by transthoracic echocardiography and graded as None/Trace (0), Mild (1+), Moderate (2+), Moderately Severe (3+), or Severe (4+)
Time Frame: 6 months postprocedure
Population: Participants with an echocardiogram evaluable for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 15
Participants
  0 | 5
  1+ | 6
  2+ | 4
  3+ | 0
  4+ | 0

3. Secondary Outcome: Implant Procedure Success
Description: Success is defined as the absence of specified adverse events evaluated through discharge following the procedure: - Aortic annular dissection, rupture, or leaflet damage - Mitral valve impingement due to implant - implant dehiscence/migration into aorta - implant dehiscence/migration into left ventricle - Hemodynamics requiring intervention - Other adverse event resulting in reoperation, explantation, or permanent disability.
Time Frame: discharge or 14 days postprocedure, whichever comes first
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 16
percentage of participants | 100 [79.4 to 100]

4. Secondary Outcome: Actuarial Freedom From Clinical Cardiovascular Events
Description: Freedom from specified clinical cardiovascular events 6 months postprocedure: - Device-related mortality - Complete heart block - Structural device failure - Endocarditis - Periprosthetic leak or dehiscence - Thromboembolism - Bleeding Event - Native Valve Deterioration - Valve Thrombosis - Hemolysis - Reoperation and explant at 6 months
Time Frame: 6 months postprocedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 16
percentage of participants | 87.5 [58.6 to 96.7]

5. Secondary Outcome: Actuarial Freedom From Clinical Cardiovascular Events
Description: as for outcome 4
Time Frame: 2 years postprocedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 16
percentage of participants | 81.2 [52.5 to 93.5]

6. Secondary Outcome: Survival Defined as Survival Free From All Cause Death at 2 Years Postprocedure.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 16
percentage of participants | 100 [79.4 to 100]

7. Secondary Outcome: Aortic Insufficiency (AI) at 2 Years
Description: Aortic insufficiency assessed by transthoracic echocardiography and graded as None/Trace (0), Mild (1+), Moderate (2+), Moderate-to-Severe (3+), or Severe (4+)
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 14
Participants
  0 | 2
  1+ | 11
  2+ | 1
  3+ | 0
  4+ | 0

8. Secondary Outcome: New York Heart Association (NYHA) Functional Capacity Classification
Description: Four classes describing the effect of cardiac disease on physical activity: Class I - disease does not limit activity; Class II - slight limitation; Class III - marked limitation; Class IV - inability to carry out any physical activity without discomfort
Time Frame: 6 months postprocedure
Population: Participants with an evaluation of this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 15
Participants
  I | 15
  II | 0
  III | 0
  IV | 0

9. Secondary Outcome: NYHA Functional Capacity Classification
Description: as for outcome 8
Time Frame: 2 years postprocedure
Population: Participants with an evaluation of this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 14
Participants
  I | 14
  II | 0
  III | 0
  IV | 0

10. Secondary Outcome: Peak Gradient - Change From Baseline
Description: Transthoracic echocardiography parameter
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 12
mm Hg | 1.1 (22.4)

11. Secondary Outcome: Peak Gradient - Change From Baseline
Description: Transthoracic echocardiography parameter
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 11
mm Hg | 1.4 (16.3)

12. Secondary Outcome: Mean Gradient - Change From Baseline
Description: Transthoracic echocardiography parameter
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 12
mm Hg | 1.2 (13.3)

13. Secondary Outcome: Mean Gradient - Change From Baseline
Description: Transthoracic echocardiography parameter
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 11
mm Hg | 2.4 (8.8)

14. Secondary Outcome: Left Ventricular (LV) Mass - Change From Baseline
Description: Left ventricular mass. Transthoracic echocardiography parameter.
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 10
g | -53.98 (76.21)

15. Secondary Outcome: LV Mass - Change From Baseline
Description: Left ventricular mass. Transthoracic echocardiography parameter.
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 10
g | -78.84 (88.00)

16. Secondary Outcome: Left Ventricular Internal Dimension (LVID) Diastole - Change From Baseline
Description: Left ventricular internal dimension. Transthoracic echocardiography parameter.
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 10
cm | -0.306 (0.843)

17. Secondary Outcome: LVID Diastole - Change From Baseline
Description: Left ventricular internal dimension. Transthoracic echocardiography parameter.
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 10
cm | -0.455 (1.023)

18. Secondary Outcome: LVID Systole - Change From Baseline
Description: Left ventricular internal dimension. Transthoracic echocardiography parameter.
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Error); unit: cm
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 8
cm | 0.030 (0.531)

19. Secondary Outcome: LVID Systole - Change From Baseline
Description: Left ventricular internal dimension. Transthoracic echocardiography parameter.
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 4
cm | -0.700 (1.108)

20. Secondary Outcome: LV Diastolic Volume - Change From Baseline
Description: Left ventricular diastolic volume. Transthoracic echocardiography parameter.
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 6
ml | 2.8 (41.3)

21. Secondary Outcome: LV Diastolic Volume - Change From Baseline
Description: Left ventricular diastolic volume. Transthoracic echocardiography parameter.
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 7
ml | 26.9 (40.9)

22. Secondary Outcome: LV Systolic Volume - Change From Baseline
Description: Left ventricular systolic volume. Transthoracic echocardiography parameter.
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 6
ml | 1.3 (25.8)

23. Secondary Outcome: LV Systolic Volume - Change From Baseline
Description: Left ventricular systolic volume. Transthoracic echocardiography parameter.
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 7
ml | 7.9 (24.9)

24. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF) - Change From Baseline
Description: Left ventricular ejection fraction. Transthoracic echocardiography parameter.
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: percentage of blood volume
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 6
percentage of blood volume | 0.00 (8.83)

25. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF) - Change From Baseline
Description: Left ventricular ejection fraction. Transthoracic echocardiography parameter.
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: percentage of blood volume
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 7
percentage of blood volume | 4.21 (10.02)

26. Secondary Outcome: Cardiac Output - Change From Baseline
Description: Stroke volume x heart rate. Transthoracic echocardiography parameter.
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 9
l/min | -0.932 (2.979)

27. Secondary Outcome: Cardiac Output - Change From Baseline
Description: Stroke volume x heart rate. Transthoracic echocardiography parameter.
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 8
l/min | -2.145 (2.679)

28. Secondary Outcome: Cardiac Index - Change From Baseline
Description: Hemodynamic parameter computed as cardiac output divided by body surface area
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: l/min/m^2
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 9
l/min/m^2 | -0.50 (1.50)

29. Secondary Outcome: Cardiac Index - Change From Baseline
Description: Hemodynamic parameter computed as cardiac output divided by body surface area
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: l/min/m^2
Arm/Group | Aortic Valve Repair
Number analyzed (Participants) | 8
l/min/m^2 | -1.09 (1.28)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Aortic Valve Repair
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 8/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aortic Valve Repair (N=16)
Aortic vlave incompetence (Cardiac disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Chronic lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aortic Valve Repair (N=16)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Pericardial effusion (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Impaired healing (General disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Laboratory test abnormal (Investigations) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic dilation (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 2 (2)
Haemorrhage (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication by the investigator was not allowed until completion of the trial. All proposed publications must be cleared by unanimous vote of a publication committee consisting of the sponsor and representatives of the study investigators. Publication materials must be submitted for review at least 60 day in advance of publication. The Sponsor may embargo publication for 60 additional days to allow for patent filing or may prevent publication if filling of such application would be premature.